CLINICAL TRIAL: NCT07181460
Title: The Effect of Exercise on Sleep Quality in Elderly Individuals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Elif Develi, Physiotherapist, Yeditepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IrmakS
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Sleep Quality
Keywords: Sleep Quality; Elderly; Exercises; Telerehabilitation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Study Group (Experimental): The sample size was determined as 18 elderly individuals.
  Interventions: Other: Exercises Program

INTERVENTIONS:
Other: Exercises Program — A program of low-intensity, safe, and functional movements was designed for older adults. It included a warm-up, breathing exercises, chair exercises, strength and mobility exercises, balance exercises, stretching, and a cool-down.

SUMMARY:
The primary objective of this study was to examine the effects of regular exercise on sleep quality in older adults. The study will assess changes in sleep quality resulting from a structured exercise program using objective and subjective measurement tools.

DETAILED DESCRIPTION:
The sample size of this study consists of a total of 18 (female and male) individuals selected in accordance with the specified inclusion and exclusion criteria.

The Sociodemographic Patient Information Form, Pittsburgh Sleep Quality Index (PSQI), SF-12/Short Form-12 Health Survey, Modified Medical Research Council Dyspnea Scale, Timed Up and Go Test, and 6-Minute Walk Test will be evaluated at the Kadıköy Municipality Living Center. All evaluations will be collected at the beginning of the study and at the end of the 16th week. Our online exercises will continue for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years of age or older,
* Being a resident of the Kadıköy Municipality Social Life House,
* Being able to independently carry out daily living activities,
* Not having any serious cardiopulmonary, neurological, or orthopedic health problems that would prevent exercise,
* Being willing to participate in the study and providing written consent,
* Being at a level where cognitive status does not prevent participation in exercise.

Exclusion Criteria:

* Those with serious cardiopulmonary, neurological, or orthopedic diseases,
* Individuals who exercise regularly,
* Individuals who did not complete the study process.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | 16 weeks
  The PSQI is a 19-item self-report measure widely used in clinical and research settings that measures sleep quality and sleep-related disturbances based on self-report over a one-month period.
SF-12 / Short Form-12 Health Survey | 16 weeks
  The SF-12 is a brief, validated health status scale derived from the SF-36 and enhanced to reproduce physical and mental component summary scores with 12 questions to reduce response burden for group comparisons.
Modified Medical Research Council (mMRC) Dyspnea Scale | 16 weeks
  The mMRC is a brief, five-point self-assessment scale from 0 to 4 that rates the impact of breathlessness on daily activities and is commonly used to classify symptom severity in respiratory diseases such as COPD.
Timed Up and Go (TUG) Test | 16 weeks
  The TUG test is described as a rapid way to quantify baseline functional mobility and fall risk in which the time it takes for the patient to get up from a chair, walk 3 meters, turn, and sit down again is measured chronometrically.
6-Minute Walk Test (6MWT) | 16 weeks
  The 6MWT is a submaximal exercise capacity test that measures the total distance a patient walks in 6 minutes; detailed guidelines for its application, safety, evaluation, and interpretation have been published by the American Thoracic Society.

CONTACTS AND LOCATIONS:
Overall Officials: Feryal Subaşı, Principal Investigator — Yeditepe University; Dilara Karaoğlu, Study Director — Yeditepe University; Deniz Aslan, MSc, Study Chair — Yeditepe University; Irmak Sıla Çetinel, Study Chair — Yeditepe University
Locations (1):
- Yeditepe University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No